CLINICAL TRIAL: NCT01783145
Title: Shared Care Follow-up After Chemotherapy for Testicular Cancer
Acronym: SCFU-TC
Status: Active, not recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: SCFU-TC 1.2011; 38710 (Other: ABR form CCMO)
Record Dates: First submitted 2013-01-27; First posted 2013-02-04 (Estimated); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Testicular Cancer
Keywords: survivorship care; testicular cancer; shared care model
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients with disseminated TC who have finished their chemotherapy, if needed followed by surgery, and who are in complete remission and currently in active follow-up.

SUMMARY:
The aim of this study is to develop and evaluate a shared care survivorship care plan (SCP) to follow-up patients with metastatic testicular cancer after completion of chemotherapy that resulted in complete remission.

DETAILED DESCRIPTION:
Rationale: Since the introduction of cisplatin, metastatic testicular cancer (TC) has become a highly curable disease. Successfully treated TC patients have a small chance of a relapse. In case of a relapse, early treatment will improve outcome. This stresses the need for a frequent and stringent follow-up scheme. Although chemotherapy is a very effective treatment, a downside of this treatment has now become apparent: chemotherapy-related complications such as the increased risk for cardiovascular disease (CVD) and secondary malignancies. CVD can manifest during treatment, but also years or decades thereafter. We recently observed early development of cardiovascular risk factors in TC patients, clustered into the metabolic syndrome. Monitoring and treatment of cardiovascular risk factors during follow-up is important to lower the chance of developing CVD.

Since TC survivors are discharged from follow-up after 10 years, collaboration between oncologists and general practitioners (GPs), in other words shared care, will ensure monitoring of cardiovascular risk factors and timely detection and treatment of late effects (cardiovascular risk management). Survivorship care plans for cancer survivors, GPs and oncologists facilitate care for long-term survivors. The testicular cancer survivor himself is the key person, who can be empowered to participate in follow-up programs and make lifestyle adjustments to decrease the risk of late effects and improve quality of life and life expectancy. However, data are scarce on the design of an evidence based effective follow-up schedule. For childhood cancer survivors a detailed guideline has been developed that can serve as a framework for adult cancer survivor follow-up.

Objective: To examine the safety and feasibility of a shared care survivorship care plan (SCP) to follow-up patients with metastatic testicular cancer after completion of chemotherapy that resulted in complete remission.

Study population: Patients that achieved a complete remission after chemotherapy for metastatic testicular cancer who are starting with follow-up or are currently in active follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with disseminated testicular cancer;
* Complete remission after chemotherapy with or without adjunctive surgery and in active follow-up;
* Age 18 years or older;
* Started with chemotherapy after January 1st 2003;
* Written informed consent.

Exclusion Criteria:

•Mental disability

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with disseminated TC who have finished their chemotherapy, if needed followed by surgery, and who are in complete remission and currently in active follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Safety of a shared care survivorship care plan (SCP). | Monitoring of safety will be done on a continuous basis with average duration of two years per participant.
  The aim of this study is to develop and evaluate a shared care SCP to follow-up patients with disseminated TC after completion of chemotherapy. Participants in the SCP will be patients, GPs and oncologists. The SCP will be defined according to follow-up guidelines for TC patients, with a focus on disease relapse and late effects.
Feasibility of a shared care survivorship care plan (SCP). | Monitoring of feasibility will be done on a continuous basis with average duration of two years per participant.
  The aim of this study is to develop and evaluate a shared care SCP to follow-up patients with disseminated TC after completion of chemotherapy. Participants in the SCP will be patients, GPs and oncologists. The SCP will be defined according to follow-up guidelines for TC patients, with a focus on disease relapse and late effects.

SECONDARY OUTCOMES:
Satisfaction with the SCP of testicular cancer survivors, GPs and oncologists. | Up to two years.
  The satisfaction with the SCP of testicular cancer survivors, GPs and oncologists will be evaluated by using questionnaires.
Willingness to migrate from hospital care to primary care. | Up to two years.
  The willingness to migrate from hospital care to primary care will be evaluated by specifying the decisions made within the SCP and by questionnaires to patients and GPs.

CONTACTS AND LOCATIONS:
Overall Officials: J.A. Gietema, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands